CLINICAL TRIAL: NCT06202235
Title: Multifrequency Renal MR Elastography in Evaluation of Chronic Kidney Diseases: Can Shear Stiffness Evaluate Renal Fibrosis in GFR-normal Patients?
Brief Title: Multifrequency MRE in Evaluation of Chronic Kidney Diseases
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Deputy director of department of radology, Shengjing Hospital
Other Study IDs: ShengjingH-CKD
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: chronic kidney disease; kidney fibrosis; MR elastography
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Magnetic Resonance Imaging; Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD Patients: Participants with diagnosed Chronic Kidney Disease will undergo the same MRI protocol as the Healthy Volunteers, including T1-weighted imaging, T2-weighted imaging, MR Elastography (MRE), Intravoxel Incoherent Motion (IVIM), Arterial Spin Labeling (ASL), T1 mapping, Blood Oxygen Level Dependent (BOLD), and Diffusion Weighted Imaging (DWI). The renal MRI will be performed within 7 days of the renal biopsy. In addition to the imaging, these participants will have their blood creatinine, cystatin C, blood pressure etc., measured.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Healthy Volunteers: Age-matched healthy individuals with no known kidney disease will be recruited. They will undergo the same MRI protocols as the CKD patient group, to establish baseline viscoelasticity parameters for comparison with the CKD patients.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Both CKD patients and healthy volunteers will undergo a comprehensive MRI protocol, including T1-weighted imaging, T2-weighted imaging, Magnetic Resonance Elastography (MRE), Intravoxel Incoherent Motion (IVIM), Arterial Spin Labeling (ASL), T1 mapping, Blood Oxygen Level Dependent (BOLD), and Diffusion-Weighted Imaging (DWI) to evaluate liver and renal characteristics.
  For CKD patients, renal MRI will be performed within 7 days of the renal biopsy . Additionally, blood tests for creatinine and cystatin C, along with blood pressure measurements, will be collected.
  Other Names: MR elastography; Intravoxel Incoherent Motion; Arterial Spin Labeling; T1 mapping; Blood Oxygen Level Dependent

SUMMARY:
Chronic Kidney Disease (CKD) is a major public health issue, leading to high mortality and the necessity for renal replacement therapy. Kidney fibrosis, resulting from chronic damage to kidney tissue, significantly determines CKD outcomes. Kidney biopsy, the gold standard for assessing fibrosis, is invasive and limited in its ability to reflect the heterogeneous nature of fibrosis. Consequently, there is growing interest in noninvasive methods, particularly Magnetic Resonance Elastography (MRE). MRE, which evaluates tissue stiffness, has shown potential for assessing kidney fibrosis. This study aims to use multifrequency MRE to assess renal fibrosis, focusing particularly on the early stages of CKD, to enhance understanding of its progression and relationship to clinical outcomes.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is a significant public health concern, impacting approximately 10% of the global population. Annually, millions face mortality or require renal replacement therapy due to CKD progression. Kidney fibrosis, a result of chronic parenchymal damage from various glomerular and tubulointerstitial insults, is a primary determinant of outcomes. Accurately assessing the extent and severity of fibrosis is vital for diagnosis and treatment. However, Glomerular Filtration Rate (GFR) may not diminish despite the presence of renal fibrosis, often until extensive damage occurs, owing to the kidney's compensatory abilities. Additionally, GFR reductions may not solely indicate chronic damage or parenchymal fibrosis.

GFR estimates using serum markers offer only rough approximations of kidney fibrosis and can be misleading. The gold standard for assessing kidney fibrosis is a kidney biopsy. However, biopsies are invasive, with potential complications and sampling errors, as they assess less than 1% of the kidney parenchyma. Given the heterogeneous and patchy nature of fibrosis within kidneys, the efficacy of biopsies is further questioned. Serial biopsies to track fibrosis progression are also impractical.

The need for noninvasive, accurate fibrosis assessment has led to research into various imaging techniques. Emerging functional MRI sequences, such as Intravoxel Incoherent Motion (IVIM) and Arterial Spin Labeling (ASL) for perfusion, Blood Oxygen Level Dependent (BOLD) for oxygenation, and T1 mapping for tissue characterization, offer multidimensional insights into renal pathology. Among these, Magnetic Resonance Elastography (MRE) appears particularly promising for directly assessing tissue mechanical properties. MRE, combining MRI with acoustic wave assessment, quantitatively determines tissue viscoelastic properties in response to external mechanical vibration. Initially developed for liver fibrosis assessment, kidney studies have shown that MRE-determined stiffness mildly negatively correlates with CKD stages and positively with fibrosis in renal allografts and diabetic kidneys. While kidney stiffness increases with fibrosis in renal allografts, it decreases with GFR in diabetic nephropathy. In CKD progression, marked by increased fibrosis and decreased GFR, these opposing effects on renal stiffness could limit MRE's applicability in CKD patients. We hypothesize that in early-stage CKD, when GFR is normal or slightly elevated, MRE could effectively determine renal fibrosis severity. To date, no study has specifically explored renal fibrosis and stiffness correlation in early-stage CKD.

Therefore, this study aims to evaluate renal fibrosis using multifrequency 3D-MRE-derived stiffness as a surrogate marker. This involves detecting renal fibrosis prior to CKD changes, distinguishing renal fibrosis from CKD stages, and comparing renal stiffness with clinicopathological correlates in CKD patients. Additionally, we will briefly explore the complementary value of MRE alongside other functional MRI metrics (IVIM, ASL, BOLD, T1 mapping) and investigate their potential efficacy in predicting the prognosis of CKD progression.

ELIGIBILITY:
Inclusion Criteria:

(1) adults with CKD defined according to the 2024 KDIGO guidelines, with either elevated SCr or abnormal proteinuria ; and (2) renal MRI was performed within 7 days of the renal biopsy.

Exclusion criteria:

(1) genitourinary malignancy, polycystic kidney disease, renal transplantation, or acute renal failure; (2) contraindications for MRI examination; (3) poor image quality; (4) kidney deformity or severe hydronephrosis on MRI; and (5) poorly defined corticomedullary demarcation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with CKD stages 1-5 and healthy age-matched adults as controls
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
Annual rate of eGFR decline | 24 months
  Serum biochemical markers, including eGFR, will be assessed, and a multi-parametric MRI scan (including MRE, IVIM, ASL, BOLD, and T1 mapping) will be performed within 7 days to collect baseline parameters. Following this, eGFR will be monitored every 3 to 6 months for a minimum of 2 years to calculate the annual rate of eGFR decline

CONTACTS AND LOCATIONS:
Overall Officials: yu shi, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Han JH, Ahn JH, Kim JS. Magnetic resonance elastography for evaluation of renal parenchyma in chronic kidney disease: a pilot study. Radiol Med. 2020 Dec;125(12):1209-1215. doi: 10.1007/s11547-020-01210-1. Epub 2020 May 4. PMID 32367323
- [Result] Grossmann M, Tzschatzsch H, Lang ST, Guo J, Bruns A, Durr M, Hoyer BF, Grittner U, Lerchbaumer M, Nguyen Trong M, Schultz M, Hamm B, Braun J, Sack I, Marticorena Garcia SR. US Time-Harmonic Elastography for the Early Detection of Glomerulonephritis. Radiology. 2019 Sep;292(3):676-684. doi: 10.1148/radiol.2019182574. Epub 2019 Jul 9. PMID 31287390